CLINICAL TRIAL: NCT02033395
Title: A Correlation Between Hair Cortisol Levels and the Development of Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-13-0910-JZ-CTIL
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants exposed to tramautic event

SUMMARY:
This observational study follows subjects who have been exposed to a traumatic event and are at risk of developing PTSD symptoms. Participants are recruited within six hours of a traumatic event, and, starting from the recruitment session, are then examined on six set points of time within a period of thirteen months. The examinations include both biological studies of cortisol in hair, blood and saliva, and psychological examinations and questionaires that assess the development and severity of PTSD symptoms.

The novel method of sampling hair cortisol allows investigators to retroactively estimate the mean levels of blood cortisol during the tree months prior to the sampling.

The study aims at further illuminating the correlation between cortisol levels both prior and following a traumatic event, and the development and severity of PTSD symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70.
* Experienced a traumatic and were at risk (or perceived risk) of serious injury to themselves or others in their surroundings.
* Signed an informed consent form.

Exclusion Criteria:

* Age under 18 or over 70.
* Severe or complex physical injury, such as severe head trauma, massive burns or injuries that require surgery under full anesthesia.
* A personal history of Psychotic state or PTSD.
* Pregnancy
* Weight below 45 Kg or over 120 Kg.
* Hair shorter than 1.5 cm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women, age 18-70, who were examined in the ER following a traumatic event.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
PTSD diagnosis and symptom severity as measured by Clinician Administered PTSD Scale (CAPS). | 13 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel